CLINICAL TRIAL: NCT06219577
Title: Subjective and Objective Performance of Systane Complete Multi-Dose PF Versus Walgreen's Lubricant Balance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Poway Eyecare and Optometry (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JM-23-02
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Systane Complete Multi-Dose PF (Other)
  Interventions: Drug: Systane Complete Multi-Dose PF
- Walgreen's Lubricant Balance (Other)
  Interventions: Drug: Walgreen's Lubricant Balance

INTERVENTIONS:
Drug: Systane Complete Multi-Dose PF — Eyedrop
  Arms: Systane Complete Multi-Dose PF
Drug: Walgreen's Lubricant Balance — Eyedrop
  Arms: Walgreen's Lubricant Balance

SUMMARY:
Single site, prospective, double-masked, randomized-controlled, two-arm study of the dry eye symptoms as well as corneal and conjunctival staining in subjects using 2 different eyedrops. Subjects will be assessed at a screening visit, and 2 follow-up visits. Clinical evaluations will include patient questionnaire, tear-breakup time, and slit lamp exam.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Subjects who currently have mild to moderate symptoms of dry eye as defined by a screening SANDE score of 20-55 inclusive (equivalent to OSDI score of 12 -32).2
* Subjects between the ages of 18-65.
* Subjects willing to comply with the prescribed regimen and schedule of eye drops.
* Subjects willing to attend all study visits.
* Subjects willing to discontinue any current artificial tear use 24 hours prior to the baseline study visit.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Ocular anterior segment infection, inflammation, abnormality, or active disease.
* History of herpetic keratitis or ocular surgery.
* Recent (within 1 year) thermal meibomian gland expression procedure including Lipiflow, iLux, or TearCare.
* Recent (within 1 year) blepharitis debridement procedure including BlephEx.
* Screening SANDE score > 55 (equivalent to OSDI score of >32).2 This is indicative of a severe dry eye.
* Screening SANDE score < 20 (equivalent to OSDI score of <12).2 This is indicative of a clinically normal eye.
* Screening non-invasive TBUT < 2 seconds, or > 10 seconds.3
* Screening NaFl score < 3 (clinically normal eye) or > 10 (severe dry eye).4
* Pregnant or lactating.
* Current use of contact lenses.
* Any change in eye drop regimen, whether OTC or RX in the last 90 days.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashouf, OD, Principal Investigator — Scripps Poway Eyecare & Optometry
Locations (1):
- Scripps Poway Eyecare & Optometry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.2) | 39.4 (15.1) | 40.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 10 | 17 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: SANDE Questionnaire
Description: The Symptom Assessment iN Dry Eye (SANDE) questionnaire.
  Subjects are asked to place an 'X' on the line to indicate both the frequency and severity of their dry eye symptoms. Each question is scored from 0 to 100. The scores for frequency and severity are used to calculate a total score, where Total Score = square.root[Q1 * Q2].
  Higher total score on the questionnaire indicates more frequent or severe dry eye symptoms.
Time Frame: Change from baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance
Number analyzed (Participants) | 35 | 35
score | -7.2 (11.7) | -2.2 (6.0)

2. Other Pre Specified Outcome: Corneal and Conjunctival Staining
Description: Baseline corneal and conjunctival staining with sodium fluorescein and Wratten filter assessed OU using the Academy of Ophthalmology 5 quadrant scheme. Each quadrant will be graded (0-3) giving a total score (by summation) of 0-15 per eye. A higher score is a worse outcome.
Time Frame: Change from baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: score
Units Other Than Participants: eyes
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
score | -2.8 (1.8) | -0.9 (1.5)

3. Other Pre Specified Outcome: Non-invasive Tear Breakup Time
Time Frame: Change from baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance
Number analyzed (Participants) | 35 | 35
Number analyzed (eyes) | 35 | 35
seconds | 3.1 (2.9) | 2.2 (4.5)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Systane Complete Multi-Dose PF | Walgreen's Lubricant Balance
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT06219577/Prot_SAP_000.pdf